CLINICAL TRIAL: NCT06391593
Title: Double-Blind, Single and Multiple Dose Study to Determine Pharmacodynamic Markers, Pharmacokinetic Parameters, and Safety of ALTO-203 in Patients With Major Depressive Disorder
Brief Title: PD, PK, and Safety of ALTO-203 in Patients With MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTO-203-201
Record Dates: First submitted 2024-04-08; First posted 2024-04-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder; Anhedonia
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia

STUDY DESIGN:
Intervention Model Description: The study will consist of two treatment periods. The initial Single-Dose Treatment Period is a randomized, double-blind, placebo-controlled 3-way crossover design with oral administration of a single dose of ALTO-203 25 μg, ALTO-203 75 μg, and matching placebo. In the subsequent Multi-Dose Parallel-Group Treatment Period, participants will receive ALTO-203 25 μg, ALTO-203 75 μg, or matching placebo randomized 1:1:1 for a total of 28 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ALTO-203 25 μg (Experimental): Drug: ALTO-203 25 μg
  Single-Dose Treatment Period: Single Dose, ALTO-203 25 μg
  Multi-Dose Treatment Period: ALTO-203 25 μg, administered orally, once daily for 28 days
  Interventions: Drug: ALTO-203 25 μg
- ALTO-203 75 μg (Experimental): Drug: ALTO-203 75 μg
  Single-Dose Treatment Period: Single Dose, ALTO-203 75 μg
  Multi-Dose Treatment Period: ALTO-203 75 μg, administered orally, once daily for 28 days
  Interventions: Drug: ALTO-203 75 μg
- Placebo (Placebo Comparator): Drug: Placebo
  Single-Dose Treatment Period: Single Dose, Placebo
  Multi-Dose Treatment Period: Placebo, administered orally, once daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALTO-203 25 μg — Active, ALTO-203 25 μg
  Arms: ALTO-203 25 μg
Drug: ALTO-203 75 μg — Active, ALTO-203 75 μg
  Arms: ALTO-203 75 μg
Drug: Placebo — Comparator, Placebo-to-match
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine the pharmacodynamic effects of ALTO-203 in patients with MDD in a randomized, placebo-controlled, single-dose crossover treatment period. Additionally, safety, tolerability, and PK will be assessed in a subsequent randomized placebo-controlled multi-dose parallel-group treatment period of 28 days.

Participants will complete subjective response questionnaires and perform cognitive tasks during the single-dose period, in which participants will receive ALTO-203 25 μg and 75 μg, as well as placebo. During the multiple-dose period, participants will receive either ALTO-203 25 μg, 75 μg , or placebo. Safety will be assessed over the single dose and 28-day multiple dose periods.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate major depressive disorder (MDD)
* Presence of anhedonia symptoms
* Not taking antidepressant at Screening Visit 2
* Willing to comply with all study assessments and procedures

Exclusion Criteria:

* Evidence of unstable medical condition
* Diagnosed bipolar disorder, psychotic disorder, or dementia
* Concurrent use of prohibited medications
* Current moderate or severe substance use disorder
* Concurrent or recent participation in another clinical trial for mental illness involving an investigational product or device

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Single Dose Period: To evaluate pharmacodynamic measures in patients with MDD after single doses of 25 μg ALTO-203, 75 μg ALTO-203, and placebo as measured by the alertness and mood components of the Bond-Lader Visual Analog Scale (BL-VAS). | Single-Dose Treatment Period - Pre-Dose, 1.5 hours, 3 hours, and 5 hours on Day 1 at Treatments 1, 2, and 3
  The Bond-Lader Visual Analogue Scale (BL-VAS) is used to measure the effects of drugs on the participants' mood. It consists of 16 VAS measurements of different mood state. For each question, the participants will rate their feelings at the time of assessment by indicating the point on the 10 cm line which best represents their mood. Each item is scored by measuring the position relative to the left-hand end of the line. The combined domains of alertness and mood will be assessed for the primary endpoint.
Multi-Dose Period: To assess the incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] during the multi-dose treatment period for ALTO-203 25 μg and ALTO-203 75 μg as compared to placebo. | Multi-Dose Treatment Period Day 1 to Day 35
  Incidence, severity, and relatedness of TEAEs, SAEs, discontinuation due to TEAEs.

SECONDARY OUTCOMES:
Single Dose Period: To assess the incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] during the single-dose treatment period for ALTO-203 25 μg and ALTO-203 75 μg as compared to placebo. | Single-Dose Treatment Period Day 1 to Day 21
  Incidence, severity, and relatedness of TEAEs, SAEs, discontinuation due to TEAEs.
Multi-Dose Period: To understand the pharmacokinetics (PK) of multi-doses of ALTO-203 in capsule formulation | Multi-Dose Treatment Period Day 1 to Day 35
  Bioanalysis of plasma samples and observed plasma concentrations of ALTO-203 after multiple days of dosing.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Site 4058, Tucson, Arizona
  - Site 4082, Oceanside, California
  - Site 4023, Torrance, California
  - Site 4059, Clermont, Florida
  - Site 4005, Orlando, Florida
  - Site 4031, Atlanta, Georgia
  - Site 4054, Pikesville, Maryland
  - Site 4036, Las Vegas, Nevada
  - Site 4022, Marlton, New Jersey
  - Site 4134, Princeton, New Jersey
  - Site 4075, Westlake, Ohio
  - Site 4040, Austin, Texas
  - Site 4072, Houston, Texas
  - Site 4007, Clinton, Utah
  - Site 4033, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No